CLINICAL TRIAL: NCT01040117
Title: Effects of Sensori-motor Integration Balance Training on Balance Disturbances in Patients With Multiple Sclerosis
Brief Title: Sensori-motor Integration Training in Multiple Sclerosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, Prof. Smania Nicola, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FISM-2009; 2009/R/27 (Other Grant/Funding Number: Fondazione Italiana Sclerosi Multipla)
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Equilibrium; Rehabilitation; Randomized Controlled Trial; Postural instability; Sensory-motor integration
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensory-motor Integration Training (Experimental)
  Interventions: Procedure: Sensory-motor Integration Training
- Conventional neurorehabilitation (Active Comparator)
  Interventions: Procedure: Conventional neurorehabilitation treatment

INTERVENTIONS:
Procedure: Sensory-motor Integration Training — Exercises will be divided into 3 levels. 1 Starting from the patient's most stable and comfortable standing position. 2 Patient will perform a single-step simulation, shifting his/her weight from one foot to the other in a frontal direction. 3 Patient will perform rapid movements, alternating feet in many directions, progressively increasing weight shifting and decreasing the support base amplitude. In the first five sessions exercises will be performed on a stable surface. During the remaining sessions patients will perform exercises on a compliant surface. During the two training periods the patient's visual condition will be progressively changed.
  Arms: Sensory-motor Integration Training
Procedure: Conventional neurorehabilitation treatment — The treatment will be consist in active joint mobilization, muscle stretching and strengthen and motor coordination exercises. In the first part of each session the active joint mobilization will be carried out while the patient was lying on a carpet in supine, prone. The training will continue with muscle stretching and strengthen exercises performed while patient will be in supine, prone (when possible) and standing.
  Motor coordination exercises will be carried out in supine position while sitting on a bench and in the standing position with a front support or with against a wall. The patient will be required to performed a total of 10 exercises with the following sequence: 6 exercises in supine position, 2 exercises in sitting position and 2 in standing position.
  Arms: Conventional neurorehabilitation

SUMMARY:
Balance impairment is a common and very disabling disturbance in people with Multiple Sclerosis. The efficacy of pharmacotherapy in treating balance impairment in MS is poorly documented in literature. Although literature dealing with the rehabilitation of balance impairment in MS is very scant, the preliminary data reports show very promising results. The present project could have a positive impact on balance and gait ability, disability, fear of falling, risk of falls and quality of life of patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
Balance impairment is one of the primary causes of disability in people with multiple sclerosis (MS). It increases the risk of falls and contributes to the development of fear of falling (FOF), a vicious cycle that leads to a limitation in daily life activities. The imbalance could be caused by motor and sensorial deficits as well as sensory-motor integration deficits. Despite the disability that balance disorders cause, literature about its' rehabilitation is very scant. To our knowledge two studies have been published on MS balance rehabilitation. The first paper described case reports on MS balance rehabilitation using the "Bobath" approach. The second paper performed a preliminary randomized controlled study describing the effectiveness in restoring balance control and reducing risk of falling using a specific training program aimed at improving sensory-motor integration in people with MS. Considering the several limitations of this study, further trials are warranted to assess the usefulness of specific sensory-motor training on balance impairment in people with MS. The aim of this randomised controlled double blinded clinical trial is to evaluate whether a training program consisting of exercises performed under different sensory conflict conditions can lead to an improvement in postural stability in patients with MS. This in turn might lead to an improvement in walking ability, autonomy in daily life activities and quality of life in people with MS.

The study will include 80 patients (age<65 years) with a diagnosis of MS relapsing remitted according to the McDonald criteria and with an Expanded Disability Status Scale score≤6.0. Patients will be divided into 2 groups, according to a randomization design. The experimental group will undergo a specific training program aimed at increasing balance ability in several sensory conflict conditions. The training program will consist of fifteen 50-minute sessions over a 5 week period (3 sessions/week). The control group will undergo conventional neurorehabilitation treatment following the same pattern of sessions as the study group. At recruitment, after treatment (5 weeks) and in the follow-up (1 month), each patient will be tested with the following clinical and instrumental procedures: Berg Balance Scale, Activities-specific Balance Confidence Scale, Fatigue Severity Scale, Postural Transfers evaluation, Multiple Sclerosis Quality Of Life (MSQOL)-54 instrument, Sensory Organization Test, GAITRite® System and platform stabilometry.

Data will be examined at first reassessment for between group differences. Data from the second reassessment will be analysed for within group differences. Sample characteristics will be summarised using descriptive statistics. Due to the small sample size, non-parametric tests will be applied: Wilcoxon's signed ranks test for within group comparisons and the Mann-withney U test for between group comparisons, both with significance set at p=0.05. Data will be analysed using SPSS v16 software.

ELIGIBILITY:
Inclusion Criteria:

* Age < 65 years
* Expanded Disability Status Scale (EDSS) 2.0 > score < 6.0 (24)
* Mini Mental State Evaluation (MMSE) score ≥ 24
* Absence of cognitive impairment
* Absence of heart problems
* Self-reported sensation of postural instability
* Ability to maintain standing position without aids for at least 1 minute
* Ability to walk independently for at least 15 metres

Exclusion Criteria:

* Disease recurrence that worsens significantly during the 3 months prior to recruitment
* Pharmacological therapy not well defined
* Presence of vestibular disorders and/or paroxysmal vertigo
* Performance of any type of rehabilitation treatment in the month prior to recruitment
* Presence of other concurrent neurological or orthopaedic diseases involving the lower limbs and/or interfering with standing position and/or walking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Clinical assessment procedures: - Berg Balance Scale (BBS) - Activities-specific Balance Confidence Scale (ABC) Instrumental assessment procedures: - Stabilometric assessment | At recruitment, after treatment (5 weeks) and in the follow-up (1 month)

SECONDARY OUTCOMES:
Clinical evaluation - Walking evaluation - Multiple Sclerosis Quality Of Life-54 (MSQOL-54) - Fatigue Severity Scale (FSS) - Postural Transfers | At recruitment, after treatment (5 weeks) and in the follow-up (1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fiaschi, Professor, Study Chair — Department of Neurological and Visual Sciences, University of Verona, Italy
Locations (2):
- Italy (2):
  - S.S.O. di Riabilitazione dell'Ospedale Policlinico, Verona, Verona
  - Section of Clinical Neurology, Department Neurological, Neuropsychological, Morphological and Movement Sciences, University of Verona, Verona, Italy, Verona

REFERENCES:
- [Background] Smania N, Picelli A, Gandolfi M, Fiaschi A, Tinazzi M. Rehabilitation of sensorimotor integration deficits in balance impairment of patients with stroke hemiparesis: a before/after pilot study. Neurol Sci. 2008 Oct;29(5):313-9. doi: 10.1007/s10072-008-0988-0. Epub 2008 Oct 21. PMID 18941933
- [Background] Cattaneo D, Jonsdottir J. Sensory impairments in quiet standing in subjects with multiple sclerosis. Mult Scler. 2009 Jan;15(1):59-67. doi: 10.1177/1352458508096874. Epub 2008 Oct 9. PMID 18845654
- [Background] Cattaneo D, Jonsdottir J, Zocchi M, Regola A. Effects of balance exercises on people with multiple sclerosis: a pilot study. Clin Rehabil. 2007 Sep;21(9):771-81. doi: 10.1177/0269215507077602. PMID 17875557
- [Derived] Gandolfi M, Munari D, Geroin C, Gajofatto A, Benedetti MD, Midiri A, Carla F, Picelli A, Waldner A, Smania N. Sensory integration balance training in patients with multiple sclerosis: A randomized, controlled trial. Mult Scler. 2015 Oct;21(11):1453-62. doi: 10.1177/1352458514562438. Epub 2015 Jan 12. PMID 25583852
- See also: The website of the Italian Foundation of Multiple Sclerosis — http://www.aism.it/index.aspx?codpage=hp